CLINICAL TRIAL: NCT05360654
Title: Superior Capsular Reconstruction With InternalBrace for Irreparable Rotator Cuff Tears
Brief Title: Superior Capsular Reconstruction With InternalBrace Study
Acronym: SCRIB
Status: Completed | Type: Observational
Sponsor: Wrightington, Wigan and Leigh NHS Foundation Trust (Other)
Collaborators: Edge Hill University (Other); University of Central Lancashire (Other)
Responsible Party: Sponsor
Other Study IDs: SCRIB
Record Dates: First submitted 2022-02-24; First posted 2022-05-04 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Superior Capsular Reconstruction
Keywords: Irreparable Rotator Cuff Tears

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of the study is to investigate the clinical and radiological outcomes after superior capsular reconstruction with InternalBrace (SCRIB) performed for irreparable rotator cuff tears.

DETAILED DESCRIPTION:
Massive rotator cuff tears which are irreparable in adults without severe gleno-humeral joint osteoarthritis pose a challenging problem. Tendon retraction, muscle atrophy and fatty infiltration often contribute to failure of repair and poor outcomes. Re-tears following primary repairs pose similar challenges. Such rotator cuff tears can be painful and functionally limiting in active individuals. The options for treatment include joint preservation techniques like debridement and subacromial decompression, partial repair, tendon transfers, InSpace balloon insertion and patch augmentation. However, all these procedures have historically led to suboptimal outcomes when compared with complete repair. Joint sacrificing or prosthetic joint replacement options include hemi-arthroplasty and reverse shoulder arthroplasty. These are not always appropriate in young participants with minimal arthritis due to concerns regarding prosthesis failure and the potential need of multiple revision surgeries in the future.

SCR is a more recently introduced technique presenting a viable alternative in this group of participants. This was first described by Hanada et al. and subsequently popularised by Mihata et al. This technique utilises either an autograft such as fascia lata, or dermal allograft to restore the superior capsule and prevent proximal migration of the humeral head. A biomechanical study has shown that SCR restores stability in the superior direction, thereby preventing abrasion and graft failure through subacromial impingement. In a recently published multiple retrospective case series, this technique showed improved functional outcomes whilst reducing pain. A recent retrospective case series of SCR at Wrightington Hospital confirmed the safety profile of this operation. 77% of participants were noted to be pain free post-operatively and were able to return to 'normal activities'. However, there are significant methodological limitations related to such retrospective studies. These studies are either the original work of the proposer of surgery, or retrospective series. Such studies remain limited in terms of wider applicability. National Institute of Health and Care Excellence (NICE), UK, has issued guidance highlighting the limitation of quality and quantity of available evidence related to this procedure. The guidance recommends the use of SCR in context of research alone. Recent studies have raised concerns related to incidence of graft failure following SCR. It is unclear what predisposes a certain patient group to graft failure. It has been suggested that addition of an InternalBrace as an additional step during SCR surgery may improve graft healing and reduce graft re-rupture rates. This is known as superior capsular reconstruction with InternalBrace (SCRIB). The investigators propose to perform a prospective study involving clinical (standardised outcome scores) and radiological (MRI scans) outcomes following SCRIB. The Investigators propose to compare graft healing rates following SCRIB versus historical controls where SCR was performed without InternalBrace.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18 and 80 years old.
* Massive Rotator cuff tears (Patte stage 3), as visualised on the MRI Scan
* Failure of non-surgical treatment.
* Patients consenting for allograft usage
* Arthroscopic assessment identifying an irreparable tear. A rotator cuff tear is deemed irreparable if it is not possible to achieve complete cover-age of the humeral head following arthroscopic release.

Exclusion Criteria:

Pre-operative

* Patients with neurological cause of weakness
* Patients with advanced arthritis affecting the joint (Kellgren-Lawrence Grade 3 to 4)
* Fixed Humeral head superior displacement (Hamada Grade 3 to 4)

Intra-operative

- Advanced cartilage loss

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with massive rotator cuff tears that have failed surgical management and are suitable for superior capsular reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
To investigate the change in clinical outcome following SCRIB using the Oxford Shoulder Score. Score scale 0 (worst) - 48 (best). | Baseline
  The Oxford Shoulder score is a 12-item patient reported outcome measure developed to assess out-comes after shoulder surgery and provide reliable, valid, and sensitive assessments of shoulder symptoms and function. The scale consists of four pain related items and eight functional items. Higher scores correlate with a better outcome.
To investigate the change in clinical outcome following SCRIB using the Oxford Shoulder Score. Score scale 0 (worst) - 48 (best) | 6 months
  The Oxford Shoulder score is a 12-item patient reported outcome measure developed to assess out-comes after shoulder surgery and provide reliable, valid, and sensitive assessments of shoulder symptoms and function. The scale consists of four pain related items and eight functional items. Higher scores correlate with a better outcome.
To investigate the change in clinical outcome following SCRIB using the Oxford Shoulder Score. Score scale 0 (worst) - 48 (best) | 12 months
  The Oxford Shoulder score is a 12-item patient reported outcome measure developed to assess out-comes after shoulder surgery and provide reliable, valid, and sensitive assessments of shoulder symptoms and function. The scale consists of four pain related items and eight functional items. Higher scores correlate with a better outcome.

SECONDARY OUTCOMES:
To investigate the difference in clinical outcome following SCRIB using the Constant Shoulder Score. o investigate the difference in clinical outcome following SCRIB using the Constant Shoulder Score. Score scale 0 (best) - 100 (worst). | Baseline
  The Constant Shoulder Score is an 8-item investigator reported outcome measure widely accepted and commonly used to assess outcomes following shoulder treatments. There are four sub-scales; patients are asked to rate their pain (15 points) and activity levels (20 points). Next, strength (25 points) and range of movement (40 points) are measured. A higher score is indicative of higher quality function. The score has been reported as reliable, responsive, and valid in assessing the impact of shoulder treatments.
To investigate the difference in clinical outcome following SCRIB using the Constant Shoulder Score. Score scale 0 (best) - 100 (worst). | 6 months
  The Constant Shoulder Score is an 8-item investigator reported outcome measure widely accepted and commonly used to assess outcomes following shoulder treatments. There are four sub-scales; patients are asked to rate their pain (15 points) and activity levels (20 points). Next, strength (25 points) and range of movement (40 points) are measured. A higher score is indicative of higher quality function. The score has been reported as reliable, responsive, and valid in assessing the impact of shoulder treatments.
To investigate the difference in clinical outcome following SCRIB using the Constant Shoulder Score. Score scale 0 (best) - 100 (worst). | 12 months
  The Constant Shoulder Score is an 8-item investigator reported outcome measure widely accepted and commonly used to assess outcomes following shoulder treatments. There are four sub-scales; patients are asked to rate their pain (15 points) and activity levels (20 points). Next, strength (25 points) and range of movement (40 points) are measured. A higher score is indicative of higher quality function. The score has been reported as reliable, responsive, and valid in assessing the impact of shoulder treatments.
To investigate the difference in clinical outcome following SCRIB using the Subjective shoulder value: Score scale 0 (worst) - 100 (best) | Baseline
  The Subjective shoulder value is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%. Subjective shoulder value has been shown to be an easily administered, responsive and valid measure of shoulder function.
To investigate the difference in clinical outcome following SCRIB using the Subjective shoulder value: Score scale 0 (worst) - 100 (best) | 6 months
  The Subjective shoulder value is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%. Subjective shoulder value has been shown to be an easily administered, responsive and valid measure of shoulder function.
To investigate the difference in clinical outcome following SCRIB using the Subjective shoulder value: Score scale 0 (worst) - 100 (best) | 12 months
  The Subjective shoulder value is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%. Subjective shoulder value has been shown to be an easily administered, responsive and valid measure of shoulder function.
To investigate the difference in clinical outcome following SCRIB using the American Shoulder and Elbow surgeons score: Score scale 0 (worst) - 100 (best) | Baseline
  The American Shoulder and Elbow surgeons score is a 17-item, 100-point scale evaluating pain and function in shoulder disorders. A higher score indicates a lower level of disability.
To investigate the difference in clinical outcome following SCRIB using the American Shoulder and Elbow surgeons score: Score scale 0 (worst) - 100 (best) | 6 months
  The American Shoulder and Elbow surgeons score is a 17-item, 100-point scale evaluating pain and function in shoulder disorders. A higher score indicates a lower level of disability.
To investigate the difference in clinical outcome following SCRIB using the American Shoulder and Elbow surgeons score: Score scale 0 (worst) - 100 (best) | 12 months
  The American Shoulder and Elbow surgeons score is a 17-item, 100-point scale evaluating pain and function in shoulder disorders. A higher score indicates a lower level of disability.
EuroQol Quality of Life Index | Baseline
  The EQ-5D is a standardised instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status. The EQ- 5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by marking the box against the most appropriate statement in each of the 5 dimensions. The EQ VAS then records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are la-belled 'Best imaginable health state' and 'Worst imaginable health state'. This in-formation can be used as a quantitative measure of health outcome as judged by the individual respondents.
EuroQol Quality of Life Index | 6 months
  The EQ-5D is a standardised instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status. The EQ- 5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by marking the box against the most appropriate statement in each of the 5 dimensions. The EQ VAS then records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are la-belled 'Best imaginable health state' and 'Worst imaginable health state'. This in-formation can be used as a quantitative measure of health outcome as judged by the individual respondents.
EuroQol Quality of Life Index | 12 months
  The EQ-5D is a standardised instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status. The EQ- 5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by marking the box against the most appropriate statement in each of the 5 dimensions. The EQ VAS then records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are la-belled 'Best imaginable health state' and 'Worst imaginable health state'. This in-formation can be used as a quantitative measure of health outcome as judged by the individual respondents.
Visual Analouge Scale. Score scale 0 (best) - 100 (worst) | Baseline
  To investigate the difference in clinical outcome following SCRIB using the Visual Analouge Scale.
Visual Analouge Scale. Score scale 0 (best) - 100 (worst) | 6 months
  To investigate the difference in clinical outcome following SCRIB using the Visual Analouge Scale.
Visual Analouge Scale. Score scale 0 (best) - 100 (worst) | 12 months
  To investigate the difference in clinical outcome following SCRIB using the Visual Analouge Scale.
Radiological healing - historic data comparison using Magnetic Resonance Imaging | 12 months
  All patients will undergo clinical diagnostic preoperative Magnetic Resonance Imaging in the work up for rotator cuff surgery. This will be used at baseline to compare with the post-operative Magnetic Resonance Imaging scan at 1 year from surgery. The Magnetic Resonance Imaging will be performed using current standard protocols for shoulder Magnetic Resonance Imaging containing axial, coronal, and sagittal sequences. Magnetic Resonance Imaging will be reported by a Musculoskeletal consultant radiologist. Graft healing would be assessed, and any healing failures would be qualified as 'graft intact' or 'graft failed'.
Graft healing measured by Magnetic Resonance Imaging | 12 months
  To assess graft healing measured by magnetic resonance scan imaging at 12 months post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Puneet Monga, Principal Investigator — Wrightington, Wigan & Leigh Teaching Hospitals NHS Foundation Trust
Locations (1):
- Wrightington, Wigan & Leigh Teaching Hospitals NHS Foundation Trust, Wigan, United Kingdom

IPD SHARING:
Plan to Share IPD: No